CLINICAL TRIAL: NCT00975455
Title: Phase 3 Study of Hematuria Evaluation
Brief Title: Hematuria Evaluation Trial for Subjects With Microscopic or Gross Hematuria to Determine the Absence or Presence of Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Predictive Biosciences (Industry)
Responsible Party: Ellen Sheets, MD, Predictive Biosciences
Other Study IDs: PBS-002
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2009-11

CONDITIONS: Microscopic or Gross Hematuria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: urine sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects with hematuria

SUMMARY:
The purpose of the study is to evaluate subjects with gross or microscopic hematuria undergoing scheduled cystoscopy to determine the absence or presence of bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* For those subjects for whom there is no family history of bladder cancer or less than a 20 pack year history of cigarette smoking, subject must be 50 or older.
* Subject's age can be lowered to 45 or older if there is a family history of bladder cancer and/or a 20 or greater pack history of cigarette smoking.
* Subject must have an intact bladder
* Subject must be scheduled to have a cystoscopy to screen for transitional call bladder cancer due to the finding of hematuria.
* Subject must be able to provide a minimum of 25 mL of urine for study purposes.
* Urine samples must be available prior to cystoscopy, bladder biopsy, and TUR.
* Subjects must be willing to sign an Institutional Review Board approved written informed consent prior to any study related procedures being performed.

Exclusion Criteria:

* Subject had a history or current diagnosis of any basal or squamous cell cancer.
* Subject had a known diagnosis of any autoimmune disease.
* Subject had known diagnosis of HIV, HCV or HBV
* Subject had disclosed voluntarily history of or current infection with TB or other systemic disease.
* Subject is currently pregnant or lactating.
* Subject had surgery within 30 days prior to enrollment
* Subject has known allergy to benzalkonium chloride.
* Subject participated in an investigational drug or device trial within 30 days prior to enrollment.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from Urology and Oncology practices.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To establish the performance characteristics of the Predictive Biosciences Assay relative to the cystoscopy results for subjects undergoing evaluation for the referral diagnosis of gross or microscopic hematuria | Initial Visit only

SECONDARY OUTCOMES:
To establish the performance characteristics of the PB assay relative to urine cytology results for subjects undergoing evaluation for the referral diagnosis of gross or microscopic hematuria. | Initial Visit

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Atlantic Urological Associates, Daytona Beach, Florida
  - Winter Park Urology, Orlando, Florida
  - Metropolitan Urology, Jeffersonville, Indiana
  - Mayo Validation Support Services, Rochester, Minnesota
  - Coastal Urology Associates, Brick, New Jersey
  - Associates in Urology, Orange, New Jersey
  - Community Care Physicians, Albany, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - Eastern Urological Associates, Greenville, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Clinics of North Texas, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas